CLINICAL TRIAL: NCT06332365
Title: Evaluating Treatment Efficacy in Oral Lichen Planus: The Role of Salivary Biomarkers
Acronym: salivaLichen
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pia Lopez Jornet (Other)
Responsible Party: Sponsor-Investigator, Pia Lopez Jornet, Head Oral Medicine, Universidad de Murcia
Organization: Universidad de Murcia (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ID: 3938/2022
Record Dates: First submitted 2024-03-19; First posted 2024-03-27 (Actual); Last update posted 2024-03-27 (Actual); Status verified 2024-02

CONDITIONS: Oral Lichen Planus; Oral Lichen Planus Related Stress
Keywords: treatment; saliva stress; oral lichen planus
MeSH Terms: conditions — Lichen Planus, Oral | interventions — Triamcinolone; lyve1b protein, zebrafish

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Randomization: The enrolled subjects were randomly assigned to one of two treatment protocols using a computer-generated table. This method ensures impartial allocation and avoids biases in treatment selection for each patient.
  Masking: Medications were prepared and packaged in identical, sealed, and numbered envelopes by the hospital pharmacy and a clinician not involved in the subsequent phases of the study. Each sealed envelope contained the protocol assignment for individual patients and written instructions for the application of the medications. Moreover, clinicians involved in treatment evaluation at each follow-up session were blinded to the treatment assigned to each patient.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group I experimental (Experimental): Group I: Received a combination of 0.1% hyaluronic acid and 0.2% triamcinolone acetonide.
  Interventions: Combination Product: Acetonide triamcinolone 0.2% +hyaluronicacid 1%
- Group II (Active Comparator): Was treated exclusively with 0.2% triamcinolone acetonide.
  Interventions: Drug: Corticoid Acetonide triamcinolone 0.2%
- Group III (Active Comparator): Received only 0.1% hyaluronic acid.
  Interventions: Drug: Hyaluronic acid 1%

INTERVENTIONS:
Combination Product: Acetonide triamcinolone 0.2% +hyaluronicacid 1% — topical application cream form twice a day for 4 weeks
  Other Names: GroupI
  Arms: Group I experimental
Drug: Corticoid Acetonide triamcinolone 0.2% — topical application cream form twice a day for 4 weeks
  Other Names: GropupII
  Arms: Group II
Drug: Hyaluronic acid 1% — topical application cream form twice a day for 4 weeks
  Other Names: groupIII
  Arms: Group III

SUMMARY:
Lichen planus, a chronic autoimmune mucocutaneous disorder, affects 0.5% to 2.2% of diverse populations. The treatment for oral lichen planus (OLP) includes a range of options, both topical and systemic therapies. Recent research has highlighted the potential of hyaluronic acid as a drug alternative, potentially offering effective management for OLP and alleviating the discomfort of this chronic condition. The objective was to assess the impact of topical hyaluronic acid on salivary oxidative stress markers in individuals suffering from oral lichen planus

DETAILED DESCRIPTION:
Interventional (Clinical Trial) Actual Enrollment : 60 participants Allocation: Randomized Intervention Model: Parallel Assignment Masking: Double (Care Provider, Outcomes Assessor) Masking Description: The clinical outcomes were assessed by an investigator masked about the treatment modality that has been used Primary Purpose: Treatment Pain , quality of life the study on oral lichen planus, three treatment groups were established:

Group I: Received a combination of 0.1% hyaluronic acid and 0.2% triamcinolone acetonide.

Group II: Was treated solely with 0.2% triamcinolone acetonide. Group III: Received only 0.1% hyaluronic acid. These groups were designed to evaluate and compare the efficacy of different treatments in patients with oral lichen planus.

ELIGIBILITY:
Inclusion Criteria:

Patients with diagnosis oral lichen planus. Patients with no history of taking corticosteroids for the last 6 months Patients who agrees to take medication.

Exclusion Criteria:

Pregnant and lactating ladies. Patients with recent dental filling associated with the lesion or associated with recent drug administration.

Patient with uncontrolled diabetes, uncontrolled hypertension,

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-01-03 (Actual); Primary Completion 2023-12-15 (Actual); Study Completion 2024-02-19 (Actual)

PRIMARY OUTCOMES:
Pain assessment scale | 4 weeks
  visual analog scale (VAS) score 0-10 higher scores mean a worse outcome.

SECONDARY OUTCOMES:
OHIP-14 questionnaire | 4 weeks
  evaluate the oral health related quality of life score 0-56 higher scores mean a worse outcome
reduction of clinical signs measure | 4 weeks
  Thongprasom Score 5 = white striae with erosive area = 1 cm2 Score 4 = white striae with erosive area < 1 cm2 Score 3 = white striae with erosive area > 1 cm2 Score 2 = white striae with atrophic area < 1 cm2 Score 1 = mild white striae only Score 0 = no lesion normal
Salivary level of oxidative stress biomarker | 4 weeks
  Salivary level of oxidative stress biomarker Amilase; Glutation, IgA, FRAP, ADA

CONTACTS AND LOCATIONS:
Locations (1):
- Pia Lopez Jornet, Murcia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Louisy A, Humbert E, Samimi M. Oral Lichen Planus: An Update on Diagnosis and Management. Am J Clin Dermatol. 2024 Jan;25(1):35-53. doi: 10.1007/s40257-023-00814-3. Epub 2023 Sep 15. PMID 37713153
- [Result] Leong XY, Gopinath D, Syeed SM, Veettil SK, Shetty NY, Menon RK. Comparative Efficacy and Safety of Interventions for the Treatment of Oral Lichen Planus: A Systematic Review and Network Meta-Analysis. J Clin Med. 2023 Apr 7;12(8):2763. doi: 10.3390/jcm12082763. PMID 37109100